CLINICAL TRIAL: NCT01250171
Title: A Randomized, Placebo-controlled, Double-blind, Proof-of-concept Study of Intravenous Secukinumab (AIN457) or Canakinumab (ACZ885) in Dry Eye Syndrome
Brief Title: The Effects of a Single Intravenous Administration of Secukinumab (AIN457) or Canakinumab (ACZ885) in Dry Eye Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPJMR0092202
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Results first posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2012-12

CONDITIONS: Dry Eye
Keywords: Dry eye; IL17/ IL-1β; Biologic
MeSH Terms: conditions — Dry Eye Syndromes | interventions — secukinumab; canakinumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Secukinumab 10 mg/kg (Experimental): Patients received a single dose of secukinumab 10 mg/kg infused intravenously over a 2 hour period.
  Interventions: Biological: Secukinumab 10 mg/kg
- Canakinumab 10 mg/kg (Experimental): Patients received a single dose of canakinumab 10 mg/kg infused intravenously over a 2 hour period.
  Interventions: Biological: Canakinumab 10 mg/kg
- Placebo (Placebo Comparator): Patients received a single placebo infusion intravenously over a 2 hour period.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Secukinumab 10 mg/kg — Secukinumab was prepared in a sterile water solution.
  Other Names: AIN457
  Arms: Secukinumab 10 mg/kg
Biological: Canakinumab 10 mg/kg — Canakinumab was prepared in a sterile water solution.
  Other Names: ACZ885
  Arms: Canakinumab 10 mg/kg
Biological: Placebo — The placebo solution for infusion contained 5% glucose.
  Arms: Placebo

SUMMARY:
This study assessed the effects of a single intravenous dose of secukinumab (AIN457) 10 mg/kg or canakinumab (ACZ885) 10 mg/kg on the signs and symptoms of dry eye. In addition, the pharmacokinetic, pharmacodynamic, and safety profiles of secukinumab and canakinumab were assessed. Blood samples were collected for the analysis of the effect of secukinumab and canakinumab on select biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18-85 with a diagnosis of moderate to severe dry eye.
* Schirmer test without anesthesia ≥ 1 and < 10 mm wetting over 5 minutes in at least 1 eye.
* Tear break up time < 7 seconds in at least 1 eye.
* Corneal staining score ≥ 3 (National Eye Institute [NEI] grading scale).
* Conjunctival redness of ≥ 1.
* Ocular surface disease index of modest to severe.
* Ability to provide informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Hemoglobin < 10 g/dl.
* Total white blood count (WBC) outside the range of 3000-14,000/µl.
* Platelets < 100,000/µl.
* Use of ocular, periocular, or systemic steroids within 60 days prior to screening.
* Use of contact lenses or prior corneal refractive surgery in either eye.
* Requirement of eye drop use during the study.
* Anesthetic or neurotrophic corneas.
* Temporary punctal plugs.
* Recent or planned exposure to live vaccinations.
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Ora Inc, 300 Brickstone Square,, Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient randomized to the secukinumab group did not receive study drug and was not included in any of the analysis sets.
Period: Overall Study
Arm/Group | Secukinumab 10 mg/kg | Canakinumab 10 mg/kg | Placebo
Started | 26 | 22 | 24
Completed | 25 | 22 | 24
Not Completed | 1 | 0 | 0
Not completed — Administrative reasons | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 10 mg/kg | Canakinumab 10 mg/kg | Placebo | Total
Number analyzed (Participants) | 25 | 22 | 24 | 71
Age Continuous [Mean (Standard Deviation); unit: years] — One patient randomized to the secukinumab group did not receive study drug and was not included in the analysis of demographic data.
  years | 55 (13) | 54 (11) | 59 (13) | 56 (13)
Sex: Female, Male [Count of Participants; unit: Participants] — One patient randomized to the secukinumab group did not receive study drug and was not included in the analysis of demographic data.
  Participants
    Female | 18 | 17 | 18 | 53
    Male | 7 | 5 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the National Eye Institute Corneal Staining Scale (NEI-CSS) at Week 4
Description: Corneal staining was done with 2% sodium fluorescein instilled into the lower palpebral conjunctiva of each eye. Staining was assessed in 5 zones of the cornea (central plus 4 quadrants) and rated on a scale of 0 (no staining) to 3 (severe, confluent staining). A mean of the 5 zones for the study eye was calculated. A higher score indicates a drier eye. A negative change score indicates improvement in dryness.
Time Frame: Baseline to Week 4
Population: All patient population: All randomized patients that received 1 full dose of a study drug per protocol. Two patients were not included in the all patient population (1 in each drug group) as they were not dosed per protocol or they did not receive the full dose of the assigned treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Secukinumab 10 mg/kg | Canakinumab 10 mg/kg | Placebo
Number analyzed (Participants) | 24 | 21 | 24
Units on a scale | 0.23 (0.4) | 0.12 (0.5) | 0.26 (0.5)

2. Secondary Outcome: Change From Baseline on the Ora Corneal Staining Scale at Weeks 1, 4, and 8
Description: Corneal staining was done with 2% sodium fluorescein instilled into the lower palpebral conjunctiva of the study eye. Staining was assessed in 3 regions (inferior, superior, and central) of the cornea and rated on a scale of 0 (no staining) to 4 (confluent staining). A mean of the 3 zones was calculated. A higher score indicates a drier eye. A negative change score indicates improvement in dryness.
Time Frame: Baseline to Weeks 1, 4, and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Secukinumab 10 mg/kg | Canakinumab 10 mg/kg | Placebo
Number analyzed (Participants) | 24 | 21 | 24
Units on a scale
  Week 1 | 0.3 (0.6) | 0.2 (0.6) | 0.4 (0.5)
  Week 4 | 0.4 (0.6) | 0.2 (0.5) | 0.4 (0.5)
  Week 8 | 0.3 (0.5) | 0.3 (0.7) | 0.2 (0.5)

3. Secondary Outcome: Change From Baseline on the Schirmer Test at Weeks 1, 4, and 8
Description: The Schirmer test measures the production of tears. A small strip of filter paper is placed inside the lower eyelid (conjunctival sac) of each eye and the eyes are kept closed for 5 minutes. The paper is removed and the length of paper that is wet is measured as an index of tear production. The amount of tear production in the study eye was ranked on a 4 point scale: 0=Normal (≥ 15 mm wetting of the paper), 1=Mild (14-9 mm wetting of the paper), 2=Moderate (8-4 mm wetting of the paper), and 3=Severe (< 4 mm wetting of the paper). A higher score indicates a drier eye. A negative change score indicates improvement in dryness.
Time Frame: Baseline to Weeks 1, 4, and 8
Population: as for outcome 1
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Secukinumab 10 mg/kg | Canakinumab 10 mg/kg | Placebo
Number analyzed (Participants) | 24 | 21 | 24
Units on a scale
  Week 1 | -0.5 [-3 to 2] | 0.1 [-3 to 3] | 0.3 [-2 to 3]
  Week 4 | -0.1 [-3 to 2] | 0.0 [-3 to 2] | 0.1 [-2 to 2]
  Week 8 | -0.1 [-3 to 2] | 0.0 [-2 to 1] | 0.3 [-2 to 3]

4. Secondary Outcome: Change From Baseline in Tear Film Breakup Time at Weeks 1, 4, and 8
Description: Tear film breakup time was defined as the time of last blink to the appearance of the first growing micelle after instilling 5 μl of non-preserved 2% sodium fluorescein into the lower palpebral conjunctiva of the study eye. Measurement was repeated 3 times and a mean tear film breakup time calculated. A lower score indicates a drier eye. A positive change score indicates improvement in dryness.
Time Frame: Baseline to Weeks 1, 4, and 8
Population: as for outcome 1
Measure: Mean (Full Range); unit: Seconds
Arm/Group | Secukinumab 10 mg/kg | Canakinumab 10 mg/kg | Placebo
Number analyzed (Participants) | 24 | 21 | 24
Seconds
  Week1 | 0.29 [-1.5 to 2.8] | 0.21 [-0.9 to 2.2] | 0.26 [-1.2 to 4.1]
  Week 4 | 0.74 [-0.7 to 6.0] | -0.16 [-3.9 to 3.0] | 0.52 [-1.2 to 2.4]
  Week 8 | 0.62 [-0.6 to 3.9] | 0.37 [-4.0 to 2.5] | 1.15 [-1.0 to 4.8]

5. Secondary Outcome: Change From Baseline on the Conjunctival Redness Scale (Ora) at Weeks 1, 4, and 8
Description: Conjunctival redness was measured in the study eye at each visit by a masked evaluator. The evaluator compared the patient's study eye with a set of 5 reference photos showing a normal eye and eyes with various degrees of redness. Redness was scored on a scale of 0-5 with a white normal eye = 0 and an eye with the most redness = 5. A higher score indicates more redness. A negative change score indicates improvement in redness.
Time Frame: Baseline to Weeks 1, 4, and 8
Population: as for outcome 1
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Secukinumab 10 mg/kg | Canakinumab 10 mg/kg | Placebo
Number analyzed (Participants) | 24 | 21 | 24
Units on a scale
  Week 1 | 0.19 [-1.0 to 1.5] | 0.10 [-1.0 to 2.0] | 0.31 [-1.0 to 1.5]
  Week 4 | 0.15 [-1.0 to 1.5] | -0.07 [-1.0 to 1.0] | 0.31 [-1.5 to 2.0]
  Week 8 | 0.02 [-1.5 to 1.5] | -0.19 [-1.0 to 0.5] | 0.21 [-1.0 to 1.5]

6. Secondary Outcome: Change From Baseline in the Ocular Surface Disease Index (OSDI) at Weeks 1, 4, and 8
Description: The OSDI is an instrument for measuring dry eye disease severity and effect on vision-related functions. Patients were asked a series of 12 questions; patients responded to the questions in regard to both eyes. Responses ranged from 0=None of the time to 4=All of the time. OSDI was calculated as the sum of the 12 question scores x 25/number of questions answered. The total score ranged from 0-100. A higher score indicates drier eyes. A negative change score indicates improvement in dryness.
Time Frame: Baseline to Weeks 1, 4, and 8
Population: as for outcome 1
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Secukinumab 10 mg/kg | Canakinumab 10 mg/kg | Placebo
Number analyzed (Participants) | 24 | 21 | 24
Units on a scale
  Week 1 | 5.6 [-16 to 30] | 8.7 [-4 to 33] | 5.5 [-13 to 27]
  Week 4 | 4.8 [-32 to 32] | 9.9 [-21 to 27] | 4.6 [-27 to 32]
  Week 8 | 2.4 [-42 to 23] | 8.2 [-27 to 34] | 3.8 [-21 to 25]

7. Secondary Outcome: Desire for Artificial Tear Use at Day 1 and Weeks 1, 4, and 8
Description: Patients were instructed to record each occurrence of a desire for topical lubricant use in a patient diary. The percentage of patients in each of 6 categories (0-5, 6-10, 11-15, 16-20, 21-25, > 25 times) indicating the number of times a patient records a desire for artificial tear use per day was calculated at each time point. The percentage was calculated using the number of patients with any reported data on that day in the respective treatment group as the denominator.
Time Frame: Day 1 and Weeks 1, 4, and 8
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Secukinumab 10 mg/kg | Canakinumab 10 mg/kg | Placebo
Number analyzed (Participants) | 24 | 21 | 24
Percentage of patients
  Day 1, 0-5 times (n=24, 21, 24) | 46 | 50 | 57
  Day 1, 6-10 times | 18 | 15 | 9
  Day 1, 11-15 times | 0 | 0 | 0
  Day 1, 16-20 times | 0 | 0 | 0
  Day 1, 21-25 times | 0 | 0 | 0
  Day 1, > 25 times | 0 | 0 | 0
  Week 1, 0-5 times (n=24, 21, 24) | 50 | 57 | 38
  Week 1, 6-10 times | 21 | 5 | 21
  Week 1, 11-15 times | 8 | 5 | 8
  Week 1, 16-20 times | 0 | 5 | 0
  Week 1, 21-25 times | 0 | 0 | 0
  Week 1, > 25 times | 0 | 0 | 0
  Week 4, 0-5 times (n=24, 21, 24) | 38 | 43 | 50
  Week 4, 6-10 times | 8 | 10 | 8
  Week 4, 11-15 times | 21 | 4 | 4
  Week 4, 16-20 times | 5 | 0 | 8
  Week 4, 21-25 times | 0 | 0 | 0
  Week 4, > 25 times | 0 | 0 | 0
  Week 8, 0-5 times (n=16, 15, 13) | 56 | 53 | 62
  Week 8, 6-10 times | 19 | 7 | 0
  Week 8, 11-15 times | 6 | 7 | 0
  Week 8, 16-20 times | 6 | 0 | 0
  Week 8, 21-25 times | 0 | 0 | 0
  Week 8, > 25 times | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity at Weeks 1, 4, and 8
Description: Best corrected visual acuity (BCVA) was assessed in the study eye. BCVA measurements were taken in a standing position using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts at an initial testing distance specific to the test charts. The BCVA score is the number of letters read correctly by the patient. A decrease in the BCVA score indicates a worsening of vision. A positive change score indicates improvement.
Time Frame: Baseline to Weeks 1, 4, and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Secukinumab 10 mg/kg | Canakinumab 10 mg/kg | Placebo
Number analyzed (Participants) | 24 | 21 | 24
Units on a scale
  Week 1 | 0.5 (4) | 0.3 (8) | 0.9 (3)
  Week 4 | 0.1 (4) | 1.2 (4) | -0.1 (4)
  Week 8 | -0.4 (4) | 1.6 (5) | -0.7 (5)

ADVERSE EVENTS:
Arm/Group | Secukinumab 10 mg/kg | Canakinumab 10 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 3/26 | 8/22 | 4/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 10 mg/kg (N=26) | Canakinumab 10 mg/kg (N=22) | Placebo (N=24)
Acute diverticulitis (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 10 mg/kg (N=26) | Canakinumab 10 mg/kg (N=22) | Placebo (N=24)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 4 | 3
White blood cell count decreased (Investigations) | 0 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.